CLINICAL TRIAL: NCT02198144
Title: Barber-Based Intervention for Hypertension in Black Men: Follow-Up Evaluation
Brief Title: Cut Your Pressure Too: The Altadena Barbershop Blood Pressure Study, Phase 2 (Intervention Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ron Victor, Director, Hypertension Center of Excellence, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BARBER-1; R01HL080582 (NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure; African American Men; Black Men
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- barbershop-based BP measurement (Other): BP monitoring by barbershop based Barbers and BP lowering medication(s)
  Interventions: Other: barbershop-based BP measurement

INTERVENTIONS:
Other: barbershop-based BP measurement — BP Measurements and blood pressure reducing medication
  Other Names: BP measurenents at their barbershop & BP reducing medication

SUMMARY:
African American men have the highest risk of any group for early death & disability from high blood pressure (BP). Clinical investigations in Dallas, TX demonstrated that African American men with high BP are able to improve their BPs when participants agree to have their BP measured at their barbershop by their barber & also take BP reducing medication as instructed by a healthcare team that includes their doctor. The goal of this study is to bring a barbershop-based model of BP measurement, treatment & follow-up from Dallas, TX to the Southern California area. This study is the 2nd of two "Barbershop" studies at Cedars-Sinai Medical Center. The 1st study was called the "Barber-Based Intervention for Hypertension in Black Men: Baseline Data Collection." In this 2nd study at Wally's barbershop, the Investigators will enlist pharmacists to integrate the community health promotion program in barbershops into the healthcare system. Barbers are uniquely positioned to facilitate hypertension case detection & referral, pharmacists are uniquely positioned to facilitate case management. Pharmacists have extensive knowledge of BP medication & they have earned the respect of patients and physicians alike. In this intervention study, barbers will be trained to measure the BP & refer those who have already been identified as having high BP to a community pharmacist for confirmation of uncontrolled high BP & development of a BP management plan. The pharmacist will work with the customers' physicians to optimize the BP medication prescribed & with individual customers to provide a user-friendly "medical home." Pharmacists will improve the customer's access to state-of-the-art medical care, The data from this study will be used to apply for a new NIH Grant. In addition, the summarized data will be shared with key stakeholders in the local community (including barbers, patrons, local healthcare providers, local pharmacists & other community leaders) to design a larger community-partnered intervention.

Specific Aims:

Aim 1. To evaluate the impact of the new intervention model on HTN control in African American males.

Aim 2. To evaluate the cost-effectiveness of the new intervention. The investigators hypothesize that the projected cost-savings to the healthcare system in reduced heart attack & stroke care will outweigh intervention & medication costs.

DETAILED DESCRIPTION:
This study is the second of two "Barbershop" studies at Cedars-Sinai Medical Center. The first study at Wally's Barbershop in Altadena, CA was called the "Barber-Based Intervention for Hypertension in Black Men: Baseline Data Collection." Men at Wally's barbershop who were found to have high blood pressure as a participant in the first study are now being asked to participate in the second Cedars-Sinai study. During this second study the men will be asked to (1) return to Wally's barbershop to have their blood pressure measured to see how they are doing now, (2) review any medicines participants are taking, and (3) work with a health care team that includes their doctor, personal barber, and a pharmacist, to help them improve their blood pressure management. This second study is a six month long study. All men that agree to participate will allow the barber to measure their blood pressure each time they return to Wally's Barbershop for a haircut and ask their barber to call the study's pharmacist to arrange a follow-up visit in a local pharmacy. The goal of this second study is to show if a team approach, which means involvement of a barber and the pharmacist, can help make it easier for men to work with their doctor to get blood pressure under control.

ROLE MODEL STORIES (DEVELOPMENT OF HEALTH MESSAGING TOOLS) Role model posters are not intended as recruitment materials, but rather are educational tools that intend to highlight positive experiences of participation. The text of the role model stories will in no way provide statements of the effectiveness of the intervention being evaluated by the present research study. Rather, they are the main health messaging tools needed to promote completion of the program in order to achieve the experiences described. Essentially they document will be used as an intervention tool for peer-based health messaging - stories from real customers in the barbershop modeling target behaviors leading that promote continued participation in the protocol by peers with the hopes of achieving to the detection, treatment, and control of high blood pressure. The Cedars-Sinai research team will interview selected participants who are already adopters of our new program, to serve as models for their peers and write the model stories that will be displayed in the barbershop. Each story will model one specific behavior, one influencing factor, and one positive outcome. Each role model story will encourage one of two desired health behaviors of potential subjects with elevated BP: 1) ask the barber to check patients' BP with each haircut, 2) schedule a follow-up visit with the study pharmacist to get patient's blood pressure under control. Large posters in the barbershop will show the model customer, his barber, and the study pharmacist who facilitated the desired behavior change. The model's (participants) own words will be used on the poster. A signed memo of agreement will be obtained from each model to record and display their story and anyone who is pictured in the story will also sign a memo of agreement to participate. The model will approve the final draft of the poster before being displayed in the barbershop, and control of high blood pressure. The Cedars-Sinai research team will interview selected participants who are already adopters of our new program, to serve as models for their peers and write the model stories that will be displayed in the barbershop. Each story will model one specific behavior, one influencing factor, and one positive outcome. Each role model story will encourage one of two desired health behaviors of potential subjects with elevated BP: 1) ask the barber to check patient's BP with each haircut, 2) schedule a follow-up visit with the study pharmacist to get patient's blood pressure under control. Large posters in the barbershop will show the model customer, his barber, and the study pharmacist who facilitated the desired behavior change. The model's (participants) own words will be used on the poster. A signed memo of agreement will be obtained from each model to record and display their story and anyone who is pictured in the story will also sign a memo of agreement to participate. The model will approve the final draft of the poster before being displayed in the barbershop.

AME11226: The investigators are requesting an amendment to our original protocol in order to pilot test a six-month Minimal Maintenance Phase that will follow the six-month Intervention Phase. The barber will continue to monitor participants' blood pressure but the study pharmacists will limit their interaction to phone calls (vs. face-to-face visits as in the Intervention Phase). In addition, all study compensation for participants will be discontinued. The goal of discontinuing such compensation is to demonstrate that participants will continue to be proactive about controlling their blood pressure as a result of intrinsic motivation with continued social support from the barber and minimal phone follow-up with the pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older) African-American male
* Regular (unsolicited) customer of this barbershop.
* There is no upper age limit

Exclusion Criteria:

* Self-assigned race/ethnicity other than African-American/ non-Hispanic black
* Female gender

  * In barbershops that cater to African-American men, approximately 2% of the clientele are women. The female customers will not be surveyed but may be offered a free blood pressure screening.
* Age < 18

  * Children will not be surveyed because the prevalence of the condition being studied (hypertension) is low and does not justify the added logistical difficulties in obtaining informed consent. Although the population surveyed will be restricted to adult black men, the barbershop provides an excellent setting to foster blood pressure screening in children and adolescents who comprise 15-20% of the barbershop clientele. During the study period, staff may offer blood pressure screening to all children accompanied by a parent and to all adolescents.
* Language other than English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
out-of-office blood pressure | Six-months
  The six-month Intervention Phase is a final blood pressure reading by research staff in the barbershop, with a goal of < 135/85 mmHg (the recommended goal for out-of-office blood pressure).

SECONDARY OUTCOMES:
Health Questionnaire | Six Months
  interim health questionnaire will be administered to collect follow-up data and evaluate progress of participation

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Cedars-Sinai Medical Center; Jeffery Wilkins, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinail Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Victor RG, Ravenell JE, Freeman A, Leonard D, Bhat DG, Shafiq M, Knowles P, Storm JS, Adhikari E, Bibbins-Domingo K, Coxson PG, Pletcher MJ, Hannan P, Haley RW. Effectiveness of a barber-based intervention for improving hypertension control in black men: the BARBER-1 study: a cluster randomized trial. Arch Intern Med. 2011 Feb 28;171(4):342-50. doi: 10.1001/archinternmed.2010.390. Epub 2010 Oct 25. PMID 20975012
- [Result] Rader F, Elashoff RM, Niknezhad S, Victor RG. Differential treatment of hypertension by primary care providers and hypertension specialists in a barber-based intervention trial to control hypertension in Black men. Am J Cardiol. 2013 Nov 1;112(9):1421-6. doi: 10.1016/j.amjcard.2013.07.004. Epub 2013 Aug 23. PMID 23978276
- [Result] Victor RG, Ravenell JE, Freeman A, Bhat DG, Storm JS, Shafiq M, Knowles P, Hannan PJ, Haley R, Leonard D. A barber-based intervention for hypertension in African American men: design of a group randomized trial. Am Heart J. 2009 Jan;157(1):30-6. doi: 10.1016/j.ahj.2008.08.018. PMID 19081393